CLINICAL TRIAL: NCT03039270
Title: Sensitivity Absolute Risk Evaluation With and Without Sonic Activation of a Desensitizing Gel Previously to in Office Bleaching in Adults.
Brief Title: Evaluation of Sensitivity With and Without Sonic Activation of a Desensitizing Gel Before in Office Bleaching in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Amazonas (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Verônica Pereira de Lima Bertocco, Graduate student, Federal University of Amazonas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 49123715.1.0000.5020; 1.310.594 (Other: Research Ethics Committee)
Record Dates: First submitted 2017-01-28; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Dentin Sensitivity; Tooth Bleaching
Keywords: Tooth Sensitivity; Tooth Bleaching; Desensitizing agent; Sonic vibration
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: Randomized, controlled clinical trial, triple-blind, split-mouth type.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither the color evaluator nor the statistician were aware of the allocation of the hemiarcs, according to the sonic activation or not of them. In the execution of the intervention, the sonic activation was applied in sites such as marginal gingiva, premolars, palatal face of the teeth, in order to mask the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Without sonic activation) (Active Comparator): Desensitizing gel applied without sonic activation, for 10 minutes, previously to the in-office bleaching.
  Interventions: Other: Control (Without sonic activation)
- With sonic activation (SMART Device®) (Experimental): Desensitizing gel applied with sonic activation, 30 seconds per tooth, previously to the in-office bleaching.
  Interventions: Other: With sonic activation (SMART Device®)

INTERVENTIONS:
Other: With sonic activation (SMART Device®) — The operator applied a desensitizing gel containing 5% potassium nitrate and 2% sodium fluoride (Desensibilize KF 2%, FGM, SC, Brazil) on the vestibular surfaces of the participant's anterior teeth. In the sonic activation side, immediately after the gel's application, sonic activation(Smart Sonic Device, FGM, SC, Brazil) was performed for 1.5 minutes in total for side (30 seconds per tooth). After the time of 30 seconds in each of the three anterior teeth of the respective side, the gel was removed from teeth with cotton. After removal of the desensitizing gel, gingival tissues were isolated and the bleaching gel were applied.
  Other Names: Sonic vibration
  Arms: With sonic activation (SMART Device®)
Other: Control (Without sonic activation) — The operator applied a desensitizing gel containing 5% potassium nitrate and 2% sodium fluoride (Desensibilize KF 2%, FGM,SC, Brazil) on the vestibular surfaces of the participant's anterior teeth. In the side allocated for application without sonic activation, gel was kept for 10 minutes, after which it was removed from the teeth. After removal of the desensitizing gel, gingival tissues were isolated and the bleaching gel were applied.
  Arms: Control (Without sonic activation)

SUMMARY:
This randomized, controlled clinical trial, triple-blind, split-mouth type was conducted aiming to assess the absolute risk of sensitivity with and without sonic activation of a desensitizing gel previously to the in-office bleaching in adults.

DETAILED DESCRIPTION:
This clinical trial evaluated the effect of sonic activation of a desensitizing gel on the occurrence of sensitivity associated with office bleaching. For this, 31 patients had their anterior superior teeth divided into right and left, according to the sonic activation (AS) or not (SS) of the desensitizer. Prior to bleaching, a desensitizing gel containing 5% potassium nitrate and 2% sodium fluoride (Desensibilize KF2%, FGM Dental Products,SC, Brazil) was applied. Sonic activation was performed with a sonic device (Smart, FGM Dental Products, SC, Brazil) at the 170 MHz frequency. A hydrogen peroxide gel (Whiteness HP Maxx, FGM Dental Products, SC, Brazil) was used in two whitening sessions. It was also performed, evaluation of the presence of cracks in enamel, through transillumination. The color change was verified using two color scales and a spectrophotometer. The dental sensitivity was recorded through a sensitivity diary answered by the patient, in the period up to 48 hours after each bleaching session. The absolute risk of tooth sensitivity was compared using the McNemar test (= 5%). The color change was analyzed from the variation of units of scale vita (SGU) and through the value of ΔE, which were compared through Student t test (α = 5%).

ELIGIBILITY:
Inclusion Criteria:

* Patients had at least six upper anterior teeth free of caries and restorations on the vestibular surface, and at least one central or canine incisor showing A2 or darker coloration, evaluated in comparison with a visual scale of color orientated by the value of the teeth (Vita Classical, Vita-Zahnfabrik- Germany).

Exclusion Criteria:

* Users of fixed orthodontic appliances, pregnant or lactating, with the presence of severe intrinsic stains on the teeth (spots on the use of tetracycline, fluorosis and depolluted teeth), who were taking any medication with action Anti-inflammatory and antioxidant, using desensitizing dentifrice and participants with previous history of dental sensitivity or any associated pathology (bruxism, gingival recession, non-carious lesion with dentin exposure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
Absolute risk of tooth sensitivity | Throughout two bleaching sessions, in the period immediately after bleaching up to 48 hours.
  Number of patients experiencing sensitivity at least once during the two whitening sessions.

SECONDARY OUTCOMES:
Bleaching effectiveness | Measured by the difference between the baseline color and 30 days after the second bleaching session.
  Change of color of teeth after bleaching.
Intensity of pain experienced, as measured by two pain scales. | Throughout two bleaching sessions, in the period immediately after bleaching up to 48 hours.
  Intensity of pain experienced

CONTACTS AND LOCATIONS:
Overall Officials: Verônica Bertocco, Principal Investigator — Federal University of Amazonas
Locations (1):
- Faculty of Dentistry, Federal University of Amazonas, Manaus, Amazonas, Brazil

IPD SHARING:
Plan to Share IPD: No